CLINICAL TRIAL: NCT06101160
Title: Long-term Follow-up of Safety and Efficacy of OnabotulinumtoxinA for Treatment of Sialorrhea in Juvenile Cerebral Palsy
Brief Title: Botulinum Toxin Injection for Sialorrhea in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hatem Samir Shehata, Professor of Neurology, Cairo University
Other Study IDs: BTX-S-JCP
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Sialorrhea
MeSH Terms: conditions — Sialorrhea | interventions — onabotulinum toxin A; Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: onaBoNT-A — injection under ultrasonography
  Other Names: Botox

SUMMARY:
A 100 units of botulinum toxin was injected in both parotid and submandibular glands for children (2 - 12 years) with incapacitating sialorrhea in juvenile cerebral palsy patients and they are followed up for 1 year

DETAILED DESCRIPTION:
This was a prospective, longitudinal analysis with 1-year follow-up of 52 children with juvenile cerebral palsy (JCP) suffering from sialorrhea enrolled from 3 tertiary pediatric neurology rehabilitation centers (two in Cairo and one in Alexandria) and subjected to repeated BoNT-A injection.

The recruitment period was between June 30, 2021, until May 1, 2022 (the last patient follow-up ended on April 30, 2023).

Intervention: 100 units of OnabotulinumtoxinA (Botox®) were injected in the parotid and submandibular glands Follow-up visits: mo 1 post-injection (for every injection session) and every 3 months thereafter

In each visit; the following efficacy variables were assessed:

Primary outcome measures: The severity and frequency of sialorrhea evaluated by Drooling Severity Scale (DSS), and Drooling Frequency Scale (DFS) and visual-analogic ratings of familial distress (VAS-FD).

Secondary outcome measure: The carers' Global Impression of Change Scale score measured on a 7-point Likert scale from -3 (very much worse) to +3 (very much improved)

Also, adverse events were assessed in each visit

ELIGIBILITY:
Inclusion Criteria:

* Juvenile cerebral palsy with age range (4 - 12 years)
* Having severe drooling (DFS > 4)
* Signing written informed consent by the legal guardians.

Exclusion Criteria:

* Previous BoNT-A injection in the last three months
* Patients receiving systemic medicine for the treatment of sialorrhea in the last 6 weeks
* Any contraindications to treatment with BoNT

Ages: 4 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Juvenile CP patients
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Drooling Severity Scale (DSS) and the Drooling Frequency Scale (DFS) | 1 year
  Each patient was assigned a severity rank according to the following grades: 1, dry: never drools; 2, mild: only the lips are wet; 3, moderate: wet on the lips and chin; 4, severe: drools to the extent that clothing becomes damp; 5, profuse: clothing, hands, tray, and objects become wet. The frequency of drooling was also rated as 1, never drools; 2, occasional drooling; 3, frequent drooling; and 4, constant drooling. The final drooling score is the summed ranking across both scales together to make a combined drooling ranking from 2 to 9.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatem Shehata, Cairo, Egypt